CLINICAL TRIAL: NCT03453749
Title: Anti-secretory Factor as a Treatment for Adults With Severe Traumatic Head Injury
Acronym: SATSWEDEN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: New study in planning
Sponsor: Peter Siesjö (Other)
Responsible Party: Sponsor-Investigator, Peter Siesjö, Professor, Consultant, Skane University Hospital
Organization: Skane University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ethics reference: 2013/144
Record Dates: First submitted 2017-12-13; First posted 2018-03-05 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Head Trauma; Intensive Care Neurological Disorder; Edema Brain
Keywords: Traumatic brain injury; Cerebral edema; Microdialysis; Inflammatory cytokines
MeSH Terms: conditions — Craniocerebral Trauma; Brain Edema; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: 5 consecutive adult patients with severe head trauma will receive treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salovum (Other): Patients will be given Salovum 1g/kg body weight/24 hours, divided into 6 dosages and given during 5 consecutive days.
  Interventions: Dietary Supplement: Salovum

INTERVENTIONS:
Dietary Supplement: Salovum — Salovum is freeze dried egg yolk, highly enriched with anti-secretory factor. Salovum is registered as a medical food by the EU

SUMMARY:
Introduction/Background Brain swelling/brain edema can occur due to many pathologies of the brain, such as infections, ischemia and trauma.

The edema can be either primarily intra-cellular or extra-cellular. The mechanisms by which edema arise are not fully known but it is proposed that inside the damaged brain, fluid will pass over the blood-brain barrier of the vessels into the extra-cellular space. The accumulation of fluid will lead to an increase in distance between the cell and its closest capillary, which may lead to energy failure and intra-cellular edema. The extra volume of the fluid leads to increased intracranial pressure, which in turn leads to an increase in blood pressure, aggravating the edema. In addition to the physiological changes that occur, the edema will be increased by the immunological response to the tissue damage with release of pro-inflammatory cytokines that give rise to both extra- and intra-cellular edema.

Today, no treatment has been proven efficient against traumatic brain edema. AF - anti-secretory factor is a 41 kDa protein that exists in humans and most animals. It was discovered due to its ability to inhibit experimental diarrhea.

AF has been proven to have an effect on Mb Menière and glaucoma. In animal models, AF has been proven efficient in reducing increased intracranial pressure caused by trauma and virus infection in the brain.

Salovum®, an egg yolk powder enriched in AF, is registered in the European Union as a medical food.

Methods: 5 adult patients with severe traumatic brain injury will be included in the trial via next of kin consent.

Medical interventions are protocol based. The protocol includes first, second and third treatment levels.

Patients included in the trial, will receive two micro-dialysis (MD) catheters in addition to standard treatment. One catheter will be placed in a separate burr hole close to the ICP and LICOX catheter, the other MD catheter will be placed in vicinity of the damaged barin tissue.

Patients will receive Salovum® 6 hours after trial inclusion. Patient dosage is 1g/kg body weight/24 hours, divided into 6 doses and administered orally, via tubing every 4 hours for 5 consecutive days.

Objective: Primary end-point is to investigate if Salovum® has a beneficiary effect on ICP.

Secondary endpoints are to investigate if Salovum® has a beneficiary effect on treatment intensity levels (TIL), brain-oxygenation, microdialysis bio-chemistry and cytokine expression in plasma and microdialysate.

DETAILED DESCRIPTION:
MD will be analysed bedside hourly for patient management, and the remaining MD samples will be frozen in -70° C for later analysis of cytokines.

An extra blood sample will be drawn twice daily, blood will be centrifuged and plasma will be frozen in -70° C for later analysis of cytokines.

ELIGIBILITY:
Inclusion Criteria:

1. Adult of either gender between 18 and 65 years.
2. Non-penetrating, isolated severe traumatic brain injury
3. GCS >3 and GCS<9 on admission or within 48 hours after injury*
4. Admission to study hospital within 24 hours of injury*
5. No known history of allergy to egg-protein
6. Planned for intracranial pressure monitoring
7. Absence of bilaterally dilated pupils
8. CT scan with traumatic pathology that is more than an isolated epidural hematoma

   * Within 24 hours of injury (for patients with GCS < 9 on admission) or Within 24 hours of deterioration (among patients deteriorating to GCS < 9 within 48 hours of injury)

Exclusion Criteria:

1. No consent
2. Systolic blood pressure below 90 mm Hg post resuscitation
3. Epidural hematoma with no other signs of intra-cranial injury
4. Penetrating injury
5. Non-fulfillment of inclusion criteria after screening and inclusion procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
ICP | Up to 7 days
  Intracranial pressure in mm Hg

SECONDARY OUTCOMES:
PtO2 | Up to 7 days
  Brain tissue oxygenation in mm Hg
Microdialysis biochemistry | Up to 7 days
  Analysis of glucose, pyruvate and lactate from micro-dialysis fluid
Cytokine expression | Up to 7 days
  Analysis of cytokines from micro-dialysis fluid
TIL | Up to 7 days
  Treatment Intensity Level, scale 0-38

CONTACTS AND LOCATIONS:
Overall Officials: David Cederberg, Consultant, Principal Investigator — Dept of Neurosurgery, Skane University Hospital, Lund, Sweden

REFERENCES:
- [Background] Eide PK, Eidsvaag VA, Hansson HA. Antisecretory factor (AF) exerts no effects on intracranial pressure (ICP) waves and ICP in patients with idiopathic normal pressure hydrocephalus and idiopathic intracranial hypertension. J Neurol Sci. 2014 Aug 15;343(1-2):132-7. doi: 10.1016/j.jns.2014.05.054. Epub 2014 Jun 2. PMID 24928077
- [Background] Zaman S, Aamir K, Lange S, Jennische E, Silfverdal SA, Hanson LA. Antisecretory factor effectively and safely stops childhood diarrhoea: a placebo-controlled, randomised study. Acta Paediatr. 2014 Jun;103(6):659-64. doi: 10.1111/apa.12581. Epub 2014 Mar 10. PMID 24484450
- [Background] Leong SC, Narayan S, Lesser TH. Antisecretory factor-inducing therapy improves patient-reported functional levels in Meniere's disease. Ann Otol Rhinol Laryngol. 2013 Oct;122(10):619-24. PMID 24294684
- [Background] Alam NH, Ashraf H, Olesen M, Salam MA, Gyr N, Meier R. Salovum egg yolk containing antisecretory factor as an adjunct therapy in severe cholera in adult males: a pilot study. J Health Popul Nutr. 2011 Aug;29(4):297-302. doi: 10.3329/jhpn.v29i4.8443. PMID 21957667
- [Background] Ulgheri C, Paganini B, Rossi F. Antisecretory factor as a potential health-promoting molecule in man and animals. Nutr Res Rev. 2010 Dec;23(2):300-13. doi: 10.1017/S0954422410000193. Epub 2010 Aug 5. PMID 20684797
- [Background] Hanner P, Rask-Andersen H, Lange S, Jennische E. Antisecretory factor-inducing therapy improves the clinical outcome in patients with Meniere's disease. Acta Otolaryngol. 2010 Feb;130(2):223-7. doi: 10.3109/00016480903022842. PMID 19479454
- [Background] Zaman S, Mannan J, Lange S, Lonnroth I, Hanson LA. B 221, a medical food containing antisecretory factor reduces child diarrhoea: a placebo controlled trial. Acta Paediatr. 2007 Nov;96(11):1655-9. doi: 10.1111/j.1651-2227.2007.00488.x. PMID 17937690
- [Background] Laurenius A, Wangberg B, Lange S, Jennische E, Lundgren BK, Bosaeus I. Antisecretory factor counteracts secretory diarrhoea of endocrine origin. Clin Nutr. 2003 Dec;22(6):549-52. doi: 10.1016/s0261-5614(03)00057-8. PMID 14613757
- [Background] Al-Olama M, Lange S, Lonnroth I, Gatzinsky K, Jennische E. Uptake of the antisecretory factor peptide AF-16 in rat blood and cerebrospinal fluid and effects on elevated intracranial pressure. Acta Neurochir (Wien). 2015 Jan;157(1):129-37. doi: 10.1007/s00701-014-2221-7. Epub 2014 Sep 24. PMID 25248325
- [Background] Al-Olama M, Wallgren A, Andersson B, Gatzinsky K, Hultborn R, Karlsson-Parra A, Lange S, Hansson HA, Jennische E. The peptide AF-16 decreases high interstitial fluid pressure in solid tumors. Acta Oncol. 2011 Oct;50(7):1098-104. doi: 10.3109/0284186X.2011.562240. Epub 2011 Mar 4. PMID 21375367